CLINICAL TRIAL: NCT05459116
Title: Visualization of Inspiratory Effort and Respiratory Mechanics to Promote Lung- and Diaphragm Protective Ventilation
Acronym: VIREM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Research Foundation Flanders (Other); Universitaire Ziekenhuizen KU Leuven (Other); The Hospital for Sick Children (Other); University of Toronto (Other); Universiteit Antwerpen (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE1712
Record Dates: First submitted 2022-06-28; First posted 2022-07-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Muscles; Respiration, Artificial; Respiratory Function Tests
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Overall group (Experimental): Placement of a nasogastric balloon
  Interventions: Device: Placement of nasogastric balloon

INTERVENTIONS:
Device: Placement of nasogastric balloon — A nasogastric balloon catheter will be inserted after inclusion. This will be a NutriVent (Sidam S.R.L., Mirandola, Italy) for patients >40kg, and a SmartCath Esophageal pressure catheter (Vyaire/Carefusion) for patients <40kg. This placement is similar to a standard nasogastric tube placement, which is a common procedure in an ICU. Potential minor side effects include a nosebleed, sore throat and erosion of the nose where the tube is anchored. All patients will receive this intervention. When the esophageal catheter becomes displaced or is accidentally removed during the study period, it will be replaced.

SUMMARY:
This is a multicentre prospective cohort trial in adult and pediatric ICU patients. The investigators will measure the effect of a patient's inspiratory effort during mechanical ventilation on the lungs and diaphragm. The investigators will daily (for a maximum of 8 days) measure esophageal pressures with a balloon catheter to quantify inspiratory effort and respiratory muscle function, and perform daily ultrasound measurements of the diaphragm and the lungs. The investigators hypothesize that a small inspiratory effort will result in the preservation of diaphragm function and have no adverse effect on lung function.

ELIGIBILITY:
Inclusion Criteria:

* age > 28 days
* weight > 3kg
* requiring invasive mechanical ventilation
* anticipated length of ventilation > 48h

Exclusion Criteria:

* refusal of consent
* mechanical ventilation ≤ 2 weeks before inclusion
* known anatomical malformation of the diaphragm (including congenital diaphragmatic hernia)
* contra-indication to the placement of a naso-gastric esophageal balloon catheter

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Tidal esophageal pressure swing (∆Pes) - D1 | ∆Pes (average over 1 minute recording) at day 1 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D2 | ∆Pes (average over 1 minute recording) at day 2 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D3 | ∆Pes (average over 1 minute recording) at day 3 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D4 | ∆Pes (average over 1 minute recording) at day 4 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D5 | ∆Pes (average over 1 minute recording) at day 5 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D6 | ∆Pes (average over 1 minute recording) at day 6 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D7 | ∆Pes (average over 1 minute recording) at day 7 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.
Tidal esophageal pressure swing (∆Pes) - D8 | ∆Pes (average over 1 minute recording) at day 8 of mechanical ventilation
  Our primary endpoint is the amount of total inspiratory muscle activity as represented by ∆Pes, measured at least once daily during the first 8 days of mechanical ventilation.

SECONDARY OUTCOMES:
Transpulmonary driving pressure (ΔPL) - D1 | ∆PL (average over 1 minute recording) at day 1 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D2 | ∆PL (average over 1 minute recording) at day 2 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D3 | ∆PL (average over 1 minute recording) at day 3 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D4 | ∆PL (average over 1 minute recording) at day 4 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D5 | ∆PL (average over 1 minute recording) at day 5 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D6 | ∆PL (average over 1 minute recording) at day 6 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D7 | ∆PL (average over 1 minute recording) at day 7 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Transpulmonary driving pressure (ΔPL) - D8 | ∆PL (average over 1 minute recording) at day 8 of mechanical ventilation
  ∆PL is calculated as change in airway pressure minus change in esophageal pressure
Occlusion pressure (P0.1) - D1 | P0.1 (average of 3 breaths) at day 1 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D2 | P0.1 (average of 3 breaths) at day 2 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D3 | P0.1 (average of 3 breaths) at day 3 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D4 | P0.1 (average of 3 breaths) at day 4 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D5 | P0.1 (average of 3 breaths) at day 5 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D6 | P0.1 (average of 3 breaths) at day 6 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D7 | P0.1 (average of 3 breaths) at day 7 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
Occlusion pressure (P0.1) - D8 | P0.1 (average of 3 breaths) at day 8 of mechanical ventilation
  P0.1 is measured during the first 100 milliseconds of a breath
End-expiratory diaphragm thickness (DTee) - D1 | DTee (average of 3 breaths) at day 1 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D2 | DTee (average of 3 breaths) at day 2 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D3 | DTee (average of 3 breaths) at day 3 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D4 | DTee (average of 3 breaths) at day 4 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D5 | DTee (average of 3 breaths) at day 5 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D6 | DTee (average of 3 breaths) at day 6 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D7 | DTee (average of 3 breaths) at day 7 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
End-expiratory diaphragm thickness (DTee) - D8 | DTee (average of 3 breaths) at day 8 of mechanical ventilation
  Measured with ultrasound. The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D1 | DTF (average of 3 breaths) at day 1 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D2 | DTF (average of 3 breaths) at day 2 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D3 | DTF (average of 3 breaths) at day 3 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D4 | DTF (average of 3 breaths) at day 4 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D5 | DTF (average of 3 breaths) at day 5 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D6 | DTF (average of 3 breaths) at day 6 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D7 | DTF (average of 3 breaths) at day 7 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Diaphragm thickening fraction (DTF) measured with ultrasound - D8 | DTF (average of 3 breaths) at day 8 of mechanical ventilation
  DTF is calculated as (Thickness at end-inspiration [DTei] - Thickness at end-expiration [DTee])/Thickness at end-expiration [DTee] × 100.
  The ultrasound probe will be positioned perpendicular to the skin at the right zone of apposition.
Duration of mechanical ventilation | From date of intubation until the date of extubation or date of death from any cause, whichever came first, assessed up to 4 months
  Cumulative duration of mechanical ventilation in days (excluding non-invasive ventilation)
Maximal inspiratory pressure (MIP) - D1 | MIP at day 1 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D2 | MIP at day 2 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D3 | MIP at day 3 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D4 | MIP at day 4 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D5 | MIP at day 5 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D6 | MIP at day 6 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D7 | MIP at day 7 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Maximal inspiratory pressure (MIP) - D8 | MIP at day 8 of mechanical ventilation
  MIP is a measure of inspiratory function. Measured once daily during an expiratory hold (± 30 seconds)
Need for tracheal reintubation after tracheal extubation | From date of inclusion until the date of reintubation or date of hospital discharge or date of death from any cause, whichever came first, assessed up to 4 months.
Lung ultrasound scores (LUSS) - D1 | LUSS at day 1 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D2 | LUSS at day 2 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D3 | LUSS at day 3 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D4 | LUSS at day 4 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D5 | LUSS at day 5 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D6 | LUSS at day 6 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D7 | LUSS at day 7 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
Lung ultrasound scores (LUSS) - D8 | LUSS at day 8 of mechanical ventilation
  Measured once daily for the first 8 days of mechanical ventilation
ICU length of stay | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 4 months
  Duration to live discharge from the ICU
ICU mortality | From date of inclusion until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 4 months
Hospital length of stay | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 4 months
  Duration to live discharge from hospital
Duration to decease | From date of intubation until the date of death from any cause, whichever came first, assessed up to 4 months
  Cumulative time to death counting from the day of intubation
Hospital mortality | From date of inclusion until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 4 months
Presence of clinical signs of muscle weakness at ICU discharge | From date of inclusion until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 4 months
Presence of clinical signs of muscle weakness at hospital discharge | From date of inclusion until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 4 months
ICU readmission rate within 48 hours | From date of ICU discharge until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 4 months
Inspiratory muscle pressure (Pmus) - D1 | Pmus at day 1 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D2 | Pmus at day 2 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D3 | Pmus at day 3 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D4 | Pmus at day 4 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D5 | Pmus at day 5 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D6 | Pmus at day 6 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D7 | Pmus at day 7 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Inspiratory muscle pressure (Pmus) - D8 | Pmus at day 8 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D1 | ∆Pocc at day 1 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D2 | ∆Pocc at day 2 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D3 | ∆Pocc at day 3 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D4 | ∆Pocc at day 4 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D5 | ∆Pocc at day 5 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D6 | ∆Pocc at day 6 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D7 | ∆Pocc at day 7 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Occlusion pressure (∆Pocc) - D8 | ∆Pocc at day 8 of mechanical ventilation
  Measured at least once daily for the first 8 days of mechanical ventilation
Esophageal pressure-time product (PTPes) - D1 | PTPes at day 1 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D2 | PTPes at day 2 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D3 | PTPes at day 3 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D4 | PTPes at day 4 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D5 | PTPes at day 5 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D6 | PTPes at day 6 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D7 | PTPes at day 7 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Esophageal pressure-time product (PTPes) - D8 | PTPes at day 8 of mechanical ventilation
  Area under the curve (AUC) of the Pes-time plot during inspiration. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D1 | VD at day 1 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D2 | VD at day 2 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D3 | VD at day 3 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D4 | VD at day 4 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D5 | VD at day 5 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D6 | VD at day 6 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D7 | VD at day 7 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.
Dead space ventilation (VD) - D8 | VD at day 8 of mechanical ventilation
  Measured with volumetric capnography (Capnostat 5, Philips) in adults only. Measured at least once daily for the first 8 days of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schepens, M.D., Ph.D., Study Director — PICU staff member
Locations (3):
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem, Antwerp
  - University Hospital Leuven (UZL), Leuven
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No